CLINICAL TRIAL: NCT07098897
Title: To Evaluate the Effect and Safety of Telitacicept and Standard Treatment for 6months in IgA Nephropathy, Single Center, Randomized, Open Label, Comparative Study
Brief Title: To Evaluate the Effect and Safety of Telitacicept and Standard Treatment for 6months in IgA Nephropathy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Dong Sun, Head of Nephrology Department, The Affiliated Hospital of Xuzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2024-KL281-01
Record Dates: First submitted 2025-07-23; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: IgA Nephropathy (IgAN)
Keywords: Telitacicept; glomerulonephritis, iga; B-cell activating factor BAFF; a proliferation-inducing ligand APRIL; IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — telitacicept; Adrenal Cortex Hormones; Prednisolone; Methylprednisolone; Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists

STUDY DESIGN:
Intervention Model Description: Single center, Open Label, Comparative study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Target Therapy Group(TTG) (Experimental): Standard Supportive Care plus Telitacicept injected Subcutaneously 160mg/time, once a week for a total of 24 weeks Target based Drug: Telitacicept 160mg once a week for 24 weeks Other Name: RC18 Drug: Standard Supportive Care plus Low dosage of Corticosteroid(≤0.5mg/kg/d) without immunosuppressants Other Name: Prednisolone / Methylprednisolone
  Interventions: Drug: Telitacicept 160mg
- Corticosteroid Therapy Group (CTG) (Active Comparator): Standard Supportive Care plus Corticosteroid Drug: Standard Supportive Care plus Corticosteroid(≤1mg/kg/d) without immunosuppressants Other Name: Prednisolone / Methylprednisolone
  Interventions: Drug: Corticosteroid
- Supportive Care Group (SCG) (Active Comparator): Standard Supportive Care Drug: ACE Inhibitor (Treatment for proteinuria suppression and blood pressure regulation) - 2-3months before randomization Drug: ARB Inhibitor (Treatment for proteinuria suppression and blood pressure regulation) - 2-3months before randomization
  Interventions: Drug: ACE Inhibitor or Angiotensin receptor antagonist

INTERVENTIONS:
Drug: Telitacicept 160mg — Currently monoclonal antibodies, that may affect the main axis of pathogenesis of IgA nephropathy and biological therapy such as Telitacicept, provides a new treatment option and altering or depletion or modulation of Gd-IgA1 producing B cells and plasma cells. At present, Telitacicept are used for clinical treatment in IgA nephropathy patient inside China, but still clear data on safety and effect, and patient's complete remission, repeated relapse data are unclear.
  Other Names: Low Dosage Corticosteroid
  Arms: Target Therapy Group(TTG)
Drug: Corticosteroid — Standard Supportive Care plus Corticosteroid(≤1mg/kg/d) without immunosuppressants
  Other Names: Prednisolone; Methylprednisolone
  Arms: Corticosteroid Therapy Group (CTG)
Drug: ACE Inhibitor or Angiotensin receptor antagonist — Drug: ACE Inhibitor (Treatment for proteinuria suppression and blood pressure regulation) - 2-3months before randomization Drug: ARB Inhibitor (Treatment for proteinuria suppression and blood pressure regulation) - 2-3months before randomization
  Other Names: ACE inhibitors; ARB inhibitors
  Arms: Supportive Care Group (SCG)

SUMMARY:
The purpose of this clinical study is to evaluate the efficacy and safety of that test group was administered with Telitacicept in patients with IgA nephropathy. The control group will be observed for up to 6months without administration of Telitacicept.

This Single center, Randomized, Open Label, Comparative study will evaluate the effect and safety of and Standard treatment for 6months in IgA Nephropathy.

DETAILED DESCRIPTION:
IgA nephropathy is the most common primary glomerulonephritis worldwide. Immune complexes, composed of galactose-deficient IgA1 and Gd-IgA1 autoantibodies, are deposited in the mesangial area of the glomeruli where they induce complement-mediated inflammation. This may result in the reduced kidney function, which can progress to end-stage kidney disease. Treatment options are very limited. It has been reported that for urinary protein excretion that is persistently more than 1g/24h and eGFR>50ml/min/1.73m2 in IgA nephropathy, the KDIGO guidelines suggest a 6-month course of glucocorticoids. Many studies further showed that 6-month course of glucocorticoids with higher side effects and leading to discontinue of glucocorticoids course before the beneficial effect of 6months course. Currently monoclonal antibodies, that may affect the main axis of pathogenesis of IgA nephropathy and biological therapy such as Telitacicept, provides a new treatment option and altering or depletion or modulation of Gd-IgA1 producing B cells and plasma cells. At present, Telitacicept are used for clinical treatment in IgA nephropathy patient inside China, but still clear data on safety and effect, and patient's complete remission, repeated relapse data are unclear. This study is a Single center, Randomized, Open Label, Comparative study. In the study, around 60-100 patients with IgA nephropathy will be enrolled, and they will be treated with Telitacicept for 6 months on the basis of conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~75 years, regardless of gender.
* Clinical evaluation and renal biopsy diagnostic for IgA nephropathy.
* Average urinary protein excretion of 0.3~3.5g/24h on two successive examinations.
* Urine Protein to Creatinine Ratio (UPCR) >= 0.75 and <= 6 milligram per milligram (mg/mg) during screening.
* Stable and optimal dose of Angiotensin converting enzyme (ACE) inhibitor and/or angiotensin II receptor blockers (ARB) at least 8 weeks prior to screening.
* eGFR≥30 ml/min/1.73m2.
* Willingness to sign an informed consent.

Exclusion Criteria:

* • Secondary IgA nephropathy such as systemic lupus erythematosus, Henoch-Schonlein purpuric nephritis and hepatitis B-associated nephritis, etc.

  * IgA nephropathy with significant glomerulosclerosis or cortical scarring.
  * Failure to meet estimated glomerular filtration rate (eGFR) and biopsy requirement criteria.
  * Rapidly progressive nephritic syndrome.
  * Acute renal failure, including rapidly progressive IgA nephropathy.
  * Current or recent (within 30 days) exposure to high-dose of steroids or immunosuppressive therapy (CTX、MMF、CsA、FK506).
  * Cirrhosis, chronic active liver disease, and serious liver function damage.
  * History of significant gastrointestinal disorders (e.g. severe chronic diarrhea or active peptic ulcer disease).
  * Any Active systemic infection or history of serious infection within one month.
  * Other major organ system disease (e.g. serious cardiovascular diseases including congestive heart failure, chronic obstructive pulmonary disease, asthma requiring oral steroid treatment or central nervous system diseases).
  * Active tuberculosis or untreated latent TB infection.
  * Malignant hypertension that is difficult to be controlled by oral drugs.
  * Known allergy, contraindication, or intolerance to the steroids.
  * Pregnancy or breast feeding at the time of entry or unwillingness to comply with measures for contraception.
  * Malignant tumors.
  * Excessive drinking or drug abuse.
  * Mental aberrations.
  * Any condition, including any uncontrolled disease state other than IgA nephropathy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete remission of proteinuria | Baseline/3months/6months
  Proteinuria<0.3g/24h
Partial remission of proteinuria | Baseline/3months/6months
  Proteinuria decline>50%
Change from baseline to 6months in 24 Hours Urine Protein in g/24hrs | Baseline/3months/6months
  Compare the Baseline 24 Hours Urine Protein to 6month
Change from baseline to 6months in eGFR | Baseline/3months/6months
  Compare the baseline eGFR to 6months

SECONDARY OUTCOMES:
Deterioration of renal function | Baseline/3months/6months
  The longitudinal decline of eGFR, serum creatinine arises>50%, or eGFR decline>25%, or onset of end-stage renal disease or dialysis treatment.
Change From Baseline Levels in Serum Immunoglobulin A (IgA) Levels in Serum Immunoglobulin G (IgG) Levels in Serum Immunoglobulin M (IgM) | Baseline/ 3months/6months
  The change in serum levels of IgA/IgG/IgM from baseline was reported.
Change From Baseline in Serum Complement C3 and C4 Levels | Baseline/3months/6months
  The change in serum component C3 and C4 from baseline were reported.
Percentage of Participants With Clinical Significant Abnormalities in Laboratory Assessments, including Blood Pressure | Baseline/3months/6months
  Laboratory investigation included haematology, biochemistry, urinalysis and Urine sediment analysis. Clinical significance was to be decided by the investigator. The systolic and diastolic blood pressure was measured after the participants have in a rested at least 3 minutes in seated position. Clinical significance was to be decided by the investigator.
Number of Participants With a Treatment-emergent Adverse Event (TEAE) | Baseline/3months/6months
  An Adverse event (AE) was any untoward medical occurrence in a clinical study participant. TEAEs were defined, within a dosing group, as AEs that started on or after the first dose of study treatment through 30 days after the last dose of study drug.
Number of Participants Who Experienced a Serious Adverse Event (SAE) | Baseline/3months/6months
  A serious adverse event (SAE) was an adverse event/reaction that results in any of the following outcomes:
  * Death
  * Is life-threatening (participant was at immediate risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe)
  * Requires participant hospitalization (formal admission to a hospital for medical reasons) or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity (ie, there was a substantial disruption of a person's ability to carry out normal life functions)
  * Is a congenital anomaly/birth defect

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China